CLINICAL TRIAL: NCT05664698
Title: Emotion Regulation Training for Adolescents With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ER_Isaksson
Record Dates: First submitted 2022-11-24; First posted 2022-12-27 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Emotion Regulation; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: One intervention (emotion regulation training) with three randomized pre-intervention baselines at different lengths.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SKILLS-ER (Experimental): Emotion regulation training
  Interventions: Behavioral: SKILLS-ER

INTERVENTIONS:
Behavioral: SKILLS-ER — The intervention (SKILLS-ER) has been developed by the research group, and aims to increase a participant's emotion regulation capacity by targeting different stages of the emotion regulation process proposed by the extended process model of emotion, i.e. identification, selection, implementation and monitoring (Sheppes, Suri & Gross, 2015). SKILLS-ER will comprise of eight sessions and include identification and differentiation of emotions, tolerance/acceptance of emotions, education of different regulatory skills, as well as on how to select, implement and monitor strategies. Sessions will take place at the Uppsala child- and adolescent psychiatry outpatient unit and consist of activating and experiential exercises administered by a clinical psychologist. Participants will gain access to internet-delivered material, such as homework assignments in-between sessions. SKILLS-ER will be delivered individually to the participants, where their parents will be involved in some sessions.

SUMMARY:
The goal of this single-case study is to pilot and evaluate a new psychological intervention (SKILLS-ER) targeting emotion regulation in adolescents with ADHD. Participants (n=9; 13-18 years of age) and their parents will partake in the intervention consisting of a total of eight sessions.

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) results in functional impairment across several life domains and is associated with high comorbidity rates and negative long-term outcomes. For adolescents with ADHD, emotional dysregulation constitute an increasing health problem. The ability to regulate one's emotions has been suggested as a major candidate for transdiagnostic sources of risk and/or resilience. A sample of adolescents (n=9; 13-18 years of age) with ADHD and emotion dysregulation will participate in an emotion regulation intervention (SKILLS-ER) in order to evaluate feasibility, potential effectiveness and to detect mechanisms that could strengthen adaptive regulation skills. The emotion regulation programme will include eight weekly sessions, and although primarily directed towards the adolescent, parents will be invited and participate in some sessions. The researchers will apply a single-case multiple baseline design across participants with repeated measurements and pre-intervention baselines at different lengths (5, 6 and 7 weeks) to which participants are randomized. The researchers will analyze the data with a combination of visual and quantitative analyses, see study protocol and statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosis
* Self- and/or parent-rated emotion regulation difficulties, as indicated via the Emotion Questionnaire (EQ).

Exclusion Criteria:

* Intellectual disability
* Autism
* Psychosis
* Bipolar disorder
* Severe depression
* Non-stabilized medication for ADHD at intake (if on medication for ADHD)
* Other ongoing psychological treatment

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in self-ratings across baseline, intervention, post-intervention with Difficulties in Emotion Regulation Scale Short Form (DERS-SF) | Changes in DERS-SF will be investigated with weekly ratings (i.e., one time per week): before (during 5, 6 or 7 weeks depending on length of baseline), during the intervention (8 ratings during 8 weeks) and after (2 ratings during 2 weeks) SKILLS-ER
  Brief version of the Difficulties in Emotion Regulation Scale, consisting of 18 items. Main outcomes include the total summed score of the DERS-SF, as well as the summed scores of individual subscales of the DERS-SF (six in total). Items are rated on a scale of 1 (= almost never) to 5 (= almost always). Items for the emotional awareness subscale are reverse-scored. Higher scores indicate higher levels of emotion regulation difficulties.
Changes in parent-ratings across baseline, intervention, post-intervention with Difficulties in Emotion Regulation Scale Short Form (DERS-SF) | Changes in DERS-SF will be investigated with weekly ratings (i.e., one time per week): before (during 5, 6 or 7 weeks depending on length of baseline), during the intervention (8 ratings during 8 weeks) and after (2 ratings during 2 weeks) SKILLS-ER
  Brief version of the Difficulties in Emotion Regulation Scale, consisting of 18 items. Main outcomes include the total summed score of the DERS-SF, as well as the summed scores of individual subscales of the DERS-SF (six in total). Items are rated on a scale of 1 (= almost never) to 5 (= almost always). Items for the emotional awareness subscale are reverse-scored. Higher scores indicate higher levels of emotion regulation difficulties.
Changes in parental rated Target behaviors (individually defined) across baseline, intervention and post-intervention | Changes in target behaviors will be investigated with daily ratings: before (1 time per day during 5, 6 or 7 days before first week of intervention phase), during the intervention (1 time per day during 8 weeks) and after (daily during 2 weeks) SKILLS-ER
  Individually defined target behaviors associated with emotion regulation which are rated in frequency.

SECONDARY OUTCOMES:
Changes in self-ratings with Cognitive Emotion Regulation Questionnaire from baseline to post-intervention | Comparing ratings before and after intervention. 1 assessment 1 week before the baseline phase, and 1 assessment 2 weeks after the intervention SKILLS-ER
  Cognitive Emotion Regulation Questionnaire (rated by participants only), which aims to measure different cognitive emotion regulation strategies (nine in total) and consists of 18 items. Items are rated on a scale from 1 (= almost never) to 5 (= almost always). Items belonging to a particular strategy are summed together, where higher scores indicate more usage of that specific strategy.
Changes in self-ratings regarding functional impairment from baseline to post-intervention | Comparing ratings before and after intervention. 1 assessment 1 week before the baseline phase, and 1 assessment 2 weeks after the intervention SKILLS-ER
  Questionnaire on functional impairment in every-day life. Scored with 4 items on a 5-point Likert scale with higher score indicating more functional impairment.
Changes in parent-ratings regarding functional impairment from baseline to post-intervention | Comparing ratings before and after intervention. 1 assessment 1 week before the baseline phase, and 1 assessment 2 weeks after the intervention SKILLS-ER
  Questionnaire on functional impairment in every-day life. Scored with 4 items on a 5-point Likert scale with higher score indicating more functional impairment.
Changes in self-ratings with Adult ADHD Self-Report Scale Adolescent version (ASRS-A) from baseline to post-intervention | Comparing ratings before and after intervention. 1 assessment 1 week before the baseline phase, and 1 assessment 2 weeks after the intervention SKILLS-ER
  Adult ADHD Self-Report Scale Adolescent version, consisting of 18 items in total. Items are rated on a scale from 0 (=never) to 4 (=very often). Items are summed together where higher scores indicate more ADHD symptoms.
Changes in parent-ratings with Adult ADHD Self-Report Scale Adolescent version (ASRS-A) from baseline to post-intervention | Comparing ratings before and after intervention. 1 assessment 1 week before the baseline phase, and 1 assessment 2 weeks after the intervention SKILLS-ER
  Adult ADHD Self-Report Scale Adolescent version, consisting of 18 items in total. Items are rated on a scale from 0 (= never) to 4 (= very often). Items are summed together, where higher scores indicate more ADHD symptoms.
Changes in self-ratings with Spence Children's Anxiety Scale Short version (SCAS-S) from baseline to post-intervention | Comparing ratings before and after intervention. 1 assessment 1 week before the baseline phase, and 1 assessment 2 weeks after the intervention SKILLS-ER
  Spence Children's Anxiety Scale Short version (SCAS-S), consisting of 19 items in total. Items are rated on a scale from 0 (= never) to 3 (= always). The total score is the sum of all the items, where higher scores indicate more anxiety symptoms.
Changes in parent-ratings with Spence Children's Anxiety Scale (SCAS) from baseline to post-intervention | Comparing ratings before and after intervention. 1 assessment 1 week before the baseline phase, and 1 assessment 2 weeks after the intervention SKILLS-ER
  Spence Children's Anxiety Scale. Items are rated on a scale from 0 (= never) to 3 (= always). The total score is the sum of all the 39 items, where higher scores indicate more anxiety symptoms.
Changes in parent-ratings with SNAP-IV from baseline to post-intervention | Comparing ratings before and after intervention. 1 assessment 1 week before the baseline phase, and 1 assessment 2 weeks after the intervention SKILLS-ER
  The sum of the eight items on the SNAP-IV scale that measures symptoms of oppositional defiant disorder (rated by parents only). Items are rated on a scale from 0 (= not at all) to 3 (= very much), with a higher score indication more symptoms.
Self-ratings with Negative Effects Questionnaire (NEQ) | Rated at 1 time-point directly after completing the last SKILLS-ER session
  Negative Effects Questionnaire. Consists of 20 items. A higher score indicates more negative effects.
Parent-ratings with Negative Effects Questionnaire (NEQ) | Rated at 1 time-point directly after completing the last SKILLS-ER session
  Negative Effects Questionnaire. Consists of 20 items. A higher score indicates more negative effects.
Self-rated Client satisfaction | Rated at 1 time-point directly after completing the last SKILLS-ER session
  Items on client satisfaction. In total 8 questions. On 4 of these questions, items are rated on a 4-point Likert scale where higher score indicated a higher satisfaction with the intervention.
Parent-rated Client satisfaction | Rated at 1 time-point directly after completing the last SKILLS-ER session
  Items on client satisfaction. In total 8 questions. On 4 of these questions, items are rated on a 4-point Likert scale where higher score indicated a higher satisfaction with the intervention.

OTHER OUTCOMES:
Adherence to treatment programme (ratings by therapists) | During intervention phase (directly after each session)
  Therapist adherence to the treatment programme will be measured by the therapist self-ratings for each session. Items are rated on a scale from 1 (=not completed) to 3 (=completed). A higher score indicate better adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Isaksson, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheppes G, Suri G, Gross JJ. Emotion regulation and psychopathology. Annu Rev Clin Psychol. 2015;11:379-405. doi: 10.1146/annurev-clinpsy-032814-112739. Epub 2015 Jan 2. PMID 25581242

DOCUMENTS (1):
  • Study Protocol (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT05664698/Prot_000.pdf